CLINICAL TRIAL: NCT01880359
Title: A Blind Randomized Multicenter Study of Accelerated Fractionated Chemo-radiotherapy With or Without the Hypoxic Cell Radiosensitizer Nimorazole (Nimoral), Using a 15-gene Signature for Hypoxia in the Treatment of Squamous Cell Carcinoma of the Head and Neck.
Brief Title: AF CRT +/- Nimorazole in HNSCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Danish Head and Neck Cancer Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EORTC-1219; 2013-002441-12 (EudraCT Number)
Record Dates: First submitted 2013-06-12; First posted 2013-06-19 (Estimated); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Locally Advanced Head and Neck HPV Negative Squamous Cell Cancers
MeSH Terms: interventions — Cisplatin; Radiotherapy; Nimorazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiotherapy+ Cisplatin+ Placebo (Placebo Comparator): Accelerated radiotherapy (Therapeutic Planning Target Volume (PTV): 70 Gray (Gy), 6 fractions/week, 35 fractions of 2 Gy, prophylactic PTV: 54.25 Gy, 6 fractions/week, 35 fractions of 1.55 Gy) + concomitant cisplatin (weekly schedule of 40mg/m2 (delivered on day 1, 8, 15, 22, 29) Patients will receive placebo (1.2 g/m2) 90 min (+/- 30 min) prior to each radiotherapy fraction but no more than 5 times a week (If the 6th radiotherapy fraction in a week is given on a separate day from the 5th fraction of radiotherapy, no nimorazole/placebo dose is received that day. If the 6th fraction of radiotherapy is given on the same day as the 5th fraction, nimorazole/placebo is given 90 minutes before the 5th radiotherapy fraction, only).
  Interventions: Drug: Cisplatin; Radiation: Radiotherapy; Drug: Placebo
- Radiotherapy+ Cisplatin+ Nimorazole (Experimental): Accelerated radiotherapy (Therapeutic PTV: 70 Gy, 6 fractions/week, 35 fractions of 2 Gy, prophylactic PTV: 54.25 Gy, 6 fractions/week, 35 fractions of 1.55 Gy) + concomitant cisplatin (weekly schedule of 40mg/m2 (delivered on day 1, 8, 15, 22, 29) .
  Patients will receive nimorazole (1.2 g/m2) 90 min (+/- 30 min) prior to each radiotherapy fraction but no more than 5 times a week (If the 6th radiotherapy fraction in a week is given on a separate day from the 5th fraction of radiotherapy, no nimorazole/placebo dose is received that day. If the 6th fraction of radiotherapy is given on the same day as the 5th fraction, nimorazole/placebo is given 90 minutes before the 5th radiotherapy fraction, only).
  Interventions: Drug: Cisplatin; Radiation: Radiotherapy; Drug: Nimorazole

INTERVENTIONS:
Drug: Cisplatin
Radiation: Radiotherapy
Drug: Placebo
  Arms: Radiotherapy+ Cisplatin+ Placebo
Drug: Nimorazole
  Arms: Radiotherapy+ Cisplatin+ Nimorazole

SUMMARY:
The drug nimorazole belongs to a class of chemicals known as 5-nitroimidazoles. Drugs from this class are used against infection. In addition, nimorazole makes tumor cells more sensitive to radiotherapy.

Therefore, the investigators want to find out whether the addition of nimorazole to the standard treatment with radiotherapy in combination with chemotherapy with cisplatin shows activity against your type of head and neck cancer and is safe.

Furthermore the investigators will investigate if a specific examination done with your tumor tissue will help to predict whether the treatment will work or not.

To find out if the activity observed with this treatment is not caused by chance alone, the investigators need to obtain data from patients who receive this treatment and from patients who receive other treatments.

The data from these two groups of patients will be compared to see which treatment is better.

Participants will be split into 2 groups. Each group will receive different treatments. The treatment each group receives is determined by chance using a computer program. This works like flipping a coin and is called randomization. This helps to make sure that groups of patients are similar when the study starts. Neither you, your study doctor, nor the study staff can influence in which group you will be placed or which treatment you will receive.

If allocated to group 1, Patient will receive radiotherapy in combination with chemotherapy with cisplatin and nimorazole as a pill. This is considered the 'experimental' treatment.

If allocated to group 2, patient will receive radiotherapy in combination with chemotherapy with cisplatin and a so called 'placebo' as a pill. The placebo is a dummy treatment. It looks like the real one, but it is not. It contains no active ingredient/medicine.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed tumors classified as stage III-IV located in the larynx, oropharynx and hypopharynx (unknown primary should be excluded; oral cavity are not eligible)
* Human papillomavirus(HPV)/p16 negative (≤70% positively stained cells), assessed locally for tumors of the oropharynx
* Tumors of the larynx and hypopharynx regardless of the HPV status
* Histopathological diagnosis of invasive squamous cell carcinoma in the primary tumor
* World Health Organization (WHO) performance 0-2
* All Hematology and biochemical investigations, should be done within 4 weeks before randomization (maximum 6 weeks before treatment starts)
* Normal bone marrow function based on routine blood samples, i.e. neutrophils ≥ 1.0 x 109/L, platelets ≥ 75 x 109/L, hemoglobin ≥ 10.0 g/dL or 6.2 mmol/L
* Normal kidney function creatinine clearance ≥ 60ml/min, and Electrolyte balance: calcium ≤ 11.5 mg/dl or 2.9 mmol/l, magnesium ≥ 1.2 mg/dl or 0.5 mmol/l
* Normal liver function assessed by routine laboratory examinations, i.e. bilirubin < 1.5 x Upper Limit of Normal (ULN), Aspartate aminotransferase (AST)< 3 x ULN, alkaline phosphatases < 3 x ULN
* No prior or current anticancer treatment to the head and neck area (e.g. radical attempted or tumor reductive surgery, neo-adjuvant chemotherapy, Epidermal Growth Factor Receptor (EGFR) inhibitors or radiotherapy).
* Patients must be candidate for curative intent external beam chemo-radiotherapy, and must be expected to complete the treatment.
* All patients should have an oral and dental examination including preferably clinical and radiological examination. Whenever indicated, extraction of dental elements should be carried out at least 10 days before treatment start;for 1-2 (max 2) monoradicular single tooth extractions (if not continous a max of 4) without bone resection 5 days (as a minimum) are allowed.
* Radiotherapy planned to start within acceptable delay (preferably within 2 weeks and a maximum of 4 weeks from randomization).
* Radiotherapy planned to start within 8 weeks from baseline imaging tumor assessment.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before randomization in the trial
* All subjects must agree to abstain from donating blood while receiving therapy and for four weeks following discontinuation of therapy.
* All subjects must agree not to share study medication with another person and to return all unused study drug to the investigator.
* Before patient registration, written informed consent must be given according to International Conference on Harmonisation /Good Clinical Practice (ICH/GCP), and national/local regulations (including material acquisition for central testing of the hypoxic signature)

Exclusion Criteria:

* Patients who have received treatment with any investigational drug substance within 4 weeks prior to randomization;
* Current participation in any other interventional clinical study;
* Pregnant or breast-feeding female patient. Pregnancy test should be done within 72 hours from treatment start;
* Female subjects of childbearing potential (defined as a sexually mature woman who 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally post-menopausal (amenorrhoea following cancer therapy does not rule out childbearing potential) for at least 12 consecutive months (i.e. has had menses at any time in the preceding 12 consecutive months)) not willing to use adequate contraception during study and for 6 month after last dose of study drug;
* Male subjects not willing to use condoms throughout study drug therapy, and for 6 months after cessation of study therapy if their partner is of childbearing potential and has no contraception;
* Known or suspected HIV infection;
* Second malignancies in the 3 years prior to study entry with the exception of surgically cured carcinoma in situ of the cervix, in situ breast cancer, incidental finding of stage T1a or T1b prostate cancer, and basal/squamous cell carcinoma of the skin;
* Uncontrolled or chronic bacterial, fungal or viral infection;
* Known or suspected hypersensitivity to component(s) of investigational product or cisplatin contraindication;
* All indicated timelines and absolute values requested by the eligibility criteria must be adhered to. However, a maximum of +/- 10% of the reference value for laboratory parameters and a maximum of +/- 3 days for timelines may be acceptable. Discussion with EORTC Headquarters and study coordinator is encouraged.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2014-07-25 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2023-01-09 (Estimated)

PRIMARY OUTCOMES:
locoregional control rate | 9 years after first patient in

SECONDARY OUTCOMES:
Time to distant metastasis | 9 years after first patient in
Time to second cancer | 9 years after first patient in
Overall survival | 9 years after first patient in
Disease-specific free survival | 9 years after first patient in
Acute and late morbidity | 9 years after first patient in

CONTACTS AND LOCATIONS:
Overall Officials: Jens Overgaard, Study Chair — Aarhus University Hospital; Vincent Grégoire, Study Chair — Cliniques Universitaires St. Luc
Locations (19):
- Australia (3):
  - Royal Brisbane And Women's Hospital, Brisbane
  - Princess Alexandra Hospital - University Of Queensland, Brisbane
  - Royal North Shore Hospital, St Leonards
- Belgium (3):
  - Hopitaux Universitaires Bordet-Erasme - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
- France (3):
  - Centre Georges-Francois-Leclerc, Dijon
  - CHU de Tours - Hopital Bretonneau, Tours
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Charite - Universitaetsmedizin Berlin - Campus Virchow-Klinikum, Berlin
  - Ludwig-Maximilians-Universitaet Muenchen - Klinikum der Universitaet Muenchen - Campus Grosshadern, München
- Netherlands (2):
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Radboud University Medical Center Nijmegen, Nijmegen
- Poland (4):
  - Medical University Of Gdansk, Gdansk
  - The Great Poland Cancer Centre, Poznan
  - Maria Sklodowska-Curie Memorial Cancer Centre, Warsaw
  - Lower Silesian Oncology Centre, Wroclaw
- Switzerland (2):
  - Hôpitaux universitaires de Genève - HUG - site de Cluse-Roseraie, Geneva
  - UniversitaetsSpital Zurich, Zurich